CLINICAL TRIAL: NCT02014129
Title: A Phase 1 Study of LY2835219 in Japanese Patients With Advanced Cancer
Brief Title: A Study of LY2835219 in Japanese Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15154; I3Y-JE-JPBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2019-09-15

CONDITIONS: Neoplasm Metastasis; Lymphoma
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 - 100 mg Abemaciclib (Experimental): 100 milligram (mg) abemaciclib administered orally every 12 hours (Q12H) in 28 day cycles. (Cycle 1 = 32 days.) Participants remained on treatment until discontinuation criteria were met.
  Interventions: Drug: LY2835219
- Cohort 2 - 150 mg Abemaciclib (Experimental): 150 mg abemaciclib administered orally Q12H in 28 day cycles. (Cycle 1 = 32 days.) Participants remained on treatment until discontinuation criteria were met.
  Interventions: Drug: LY2835219
- Cohort 3 - 200 mg Abemaciclib (Experimental): 200 mg abemaciclib administered orally Q12H in 28 day cycles. (Cycle 1 = 32 days.) Participants remained on treatment until discontinuation criteria were met.
  Interventions: Drug: LY2835219

INTERVENTIONS:
Drug: LY2835219 — Administered orally
  Other Names: abemaciclib

SUMMARY:
The main purpose of this study is to evaluate safety and side effects of LY2835219 in Japanese participants with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of cancer (either a solid tumor or a lymphoma) that is advanced and/or metastatic
* Must be, in the judgment of the investigator, an appropriate candidate for the experimental therapy after available standard therapies have failed to provide clinical benefit for their disease
* Have the presence of measurable or non-measurable disease as defined by the Response Evaluation Criteria in Solid Tumors Guideline Version 1.1, or the Revised Response Criteria for Malignant Lymphoma Guideline
* Have adequate organ function
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, immunotherapy, and investigational therapy, for at least 21 days before the first dose of study drug and recovered from the acute effects of any such therapy
* Males must agree to use medically approved barrier contraceptive precautions during the study and for 3 months following the last dose of study drug
* Females with child bearing potential: must agree to use medically approved contraceptive precautions during the study and for 3 months following the last dose of study drug, must have had a negative serum or urine pregnancy test ≤7 days before the first dose of study drug.
* A breastfeeding woman must not be breastfeeding. If a female who stops breastfeeding enters the study, the female must stop breastfeeding from the day of the first study drug administration until at least 3 months after the last administration
* Have an estimated life expectancy of ≥12 weeks
* Are able to swallow capsules

Exclusion Criteria:

* Have received treatment within 21 days of the initial dose of study drug with an experimental agent for noncancer indications that has not received regulatory approval for any indication
* Have a medical history of any of the following conditions: presyncope or syncope of either unexplained or cardiovascular etiology, ventricular arrhythmia (e.g., ventricular tachycardia and ventricular fibrillation) or sudden cardiac arrest
* Have a baseline with any of the following findings on screening electrocardiogram (ECG): ventricular tachycardia, ventricular fibrillation, abnormal QTc using Bazett's formula (QTcB) (defined as ≥470 milliseconds), or evidence of acute myocardial ischemia
* Have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study (for example, history of major surgical resection involving the stomach or small bowel)
* Have symptomatic central nervous system (CNS) malignancy or metastasis. For asymptomatic participants without history of CNS malignancy or metastases
* Have evidence or history of a leukemia
* Have received a stem-cell transplant. As an exception, a participant with lymphoma who received an autologous stem-cell transplant is eligible for the study, if more than 75 days have passed before the initial dose of study drug
* Have active bacterial, fungal, and/or known viral infection (for example, human immunodeficiency virus [HIV], hepatitis B, or hepatitis C)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gelbert LM, Cai S, Lin X, Sanchez-Martinez C, Del Prado M, Lallena MJ, Torres R, Ajamie RT, Wishart GN, Flack RS, Neubauer BL, Young J, Chan EM, Iversen P, Cronier D, Kreklau E, de Dios A. Preclinical characterization of the CDK4/6 inhibitor LY2835219: in-vivo cell cycle-dependent/independent anti-tumor activities alone/in combination with gemcitabine. Invest New Drugs. 2014 Oct;32(5):825-37. doi: 10.1007/s10637-014-0120-7. Epub 2014 Jun 13. PMID 24919854

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants completed the trial if they received at least one dose of study drug and met discontinuation criteria.
Period: Overall Study
Arm/Group | Cohort 1 - 100 mg Abemaciclib | Cohort 2 - 150 mg Abemaciclib | Cohort 3 - 200 mg Abemaciclib
Started | 3 | 3 | 6
Received at Least One Dose of Study Drug | 3 | 3 | 6
Completed | 3 | 3 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Cohort 1 - 100 mg Abemaciclib: 100 mg abemaciclib administered orally Q12H in 28 day cycles. (Cycle 1 = 32 days.) Participants remained on treatment until discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 100 mg Abemaciclib | Cohort 2 - 150 mg Abemaciclib | Cohort 3 - 200 mg Abemaciclib | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.06) | 63.0 (1.00) | 56.0 (11.70) | 59.1 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 5 | 7
  Male | 2 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3 | 3 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abemaciclib Dose-Limiting Toxicity (DLT)
Description: DLT is defined as an adverse event between Day -3 and Day 29 of Cycle 1 that is possibly related to the study drug and fulfills any one of the following criteria using the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.
Time Frame: Cycle 1 = 32 days
Population: All participants who received at least one dose of study drug and took at least 75% of planned dose in Cycle 1 or experienced a DLT in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 100 mg Abemaciclib | Cohort 2 - 150 mg Abemaciclib | Cohort 3 - 200 mg Abemaciclib
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 1

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of Abemaciclib
Description: Maximum plasma concentration on Day -3 and Day 28 of Cycle 1.
Time Frame: Cycle 1 Day -3: Predose, 1, 2, 4, 6, 8, 10, 24, 48 and 72 hours (hr) postdose; Cycle 1 Day 28: Predose, 1, 2, 4, 6, 8, 10 and 24 hr postdose (Cycle 1 = 32 days)
Population: All participants who received at least one dose of study drug and had evaluable data for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1 - 100 mg Abemaciclib | Cohort 2 - 150 mg Abemaciclib | Cohort 3 - 200 mg Abemaciclib
Number analyzed (Participants) | 3 | 3 | 6
nanogram per milliliter (ng/mL)
  Cycle 1 Day -3 | 127 (51) | 167 (40) | 214 (87)
  Cycle 1 Day 28: number analyzed (Participants) | 2 | 2 | 5
  Cycle 1 Day 28 | NA (NA) — N=2, no geometric mean or Coefficient of variation (CV), individual values reported: 231.58, 1379.20. | NA (NA) — N=2, no geometric mean or CV, individual values reported:1381.46, 148.86. | 298 (64)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve (AUC) of Abemaciclib
Description: AUC on Day -3 and Day 28 of Cycle 1 are AUC from time zero to infinity [AUC(0-∞)] and AUC during one dosing interval at steady state (AUCτ,ss), respectively.
Time Frame: Cycle 1 Day -3: Predose, 1, 2, 4, 6, 8, 10, 24, 48 and 72 hr postdose; Cycle 1 Day 28: Predose, 1, 2, 4, 6, 8, 10 and 24 hr postdose (Cycle 1 = 32 days)
Population: All participants who received at least one dose of study drug and had evaluable data for AUC.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/Millilitre (ng*hr/mL)
Arm/Group | Cohort 1 - 100 mg Abemaciclib | Cohort 2 - 150 mg Abemaciclib | Cohort 3 - 200 mg Abemaciclib
Number analyzed (Participants) | 3 | 3 | 6
Nanogram*hour/Millilitre (ng*hr/mL)
  AUC(0-∞): number analyzed (Participants) | 2 | 3 | 6
  AUC(0-∞) | NA (NA) — N=2, no geometric mean or CV, individual values reported: 6970, 6450. | 4450 (39) | 5480 (95)
  AUCτ,ss (n=2,2,5): number analyzed (Participants) | 2 | 2 | 5
  AUCτ,ss (n=2,2,5) | NA (NA) — N=2, no geometric mean or CV, individual values reported: 2070, 14100. | NA (NA) — N=2, no geometric mean or CV, individual values reported: 15500, 1460. | 3020 (73)

4. Secondary Outcome: Percentage of Participants With a Tumor Response: Objective Response Rate (ORR)
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. Complete Response (CR) was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; Partial Response (PR) was defined as having at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: Baseline to Measured Progressive Disease (Up To 24 months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 - 100 mg Abemaciclib | Cohort 2 - 150 mg Abemaciclib | Cohort 3 - 200 mg Abemaciclib
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | Cohort 1 - 100 mg Abemaciclib | Cohort 2 - 150 mg Abemaciclib | Cohort 3 - 200 mg Abemaciclib
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 100 mg Abemaciclib (N=3) | Cohort 2 - 150 mg Abemaciclib (N=3) | Cohort 3 - 200 mg Abemaciclib (N=6)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 100 mg Abemaciclib (N=3) | Cohort 2 - 150 mg Abemaciclib (N=3) | Cohort 3 - 200 mg Abemaciclib (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (12)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 6 (8)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (6)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 2 (3)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (3)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2) | 5 (6)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (2) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (4)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 4 (6)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days